CLINICAL TRIAL: NCT06417268
Title: Ultrasound-Guided Combined Pericapsular Nerve Group Block and Lateral Femoral Cutaneous Nerve Block Versus Caudal Block for Postoperative Analgesia in Pediatric Hip Surgeries. A Randomized Controlled Study.
Brief Title: Combined Pericapsular Nerve Group Block and Lateral Femoral Cutaneous Nerve Block for Pediatric Hip Surgeries
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, maged gamal, Anesthesia lecturer, Kasr El Aini Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: MD-16-2024
Record Dates: First submitted 2024-03-20; First posted 2024-05-16 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Pericapsular Nerve Group Block
Keywords: Hip surgery; Lateral Femoral Cutaneous Nerve Block
MeSH Terms: interventions — Fentanyl; Morphine; Acetaminophen

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group C (Active Comparator): Patients will receive caudal analgesia
  Interventions: Procedure: Caudal epidural analgesia; Drug: Fentanyl; Drug: Morphine; Drug: Acetaminophen
- Group B (Active Comparator): patients will receive PENG block and Lateral Femoral Cutaneous Nerve block
  Interventions: Procedure: Ultrasound-guided Combined Pericapsular Nerve Group Block; Procedure: Ultrasound-guided Lateral Femoral Cutaneous Nerve Block; Drug: Fentanyl; Drug: Morphine; Drug: Acetaminophen

INTERVENTIONS:
Procedure: Caudal epidural analgesia — patient will be placed in the left lateral position with flexed hips.After palpating the landmarks (the upper posterior iliac spine and sacral hiatus from the edges of an equilateral triangle), an epidural puncture is performed in the most proximal region of the sacral hiatus with the needle inclined 45-60° to the skin. While palpating with the index finger of the left hand, the needle is inserted immediately below the spinous process S4.
  After perforating the membrane, the needle will be advanced no more than 1-3 mm to avoid a bloody puncture or an intrathecal injection, The confirmation of the correct position of the caudal needle before injection by performing the modified 'swoosh' test" performed by auscultation at the thoracolumbar region with a stethoscope while injecting 2 mL of saline. Bupivacaine 0.25% at a dose of 1 ml/kg will be injected, with care taken not to exceed the maximum recommended dose (2 mg/kg).
  Arms: Group C
Procedure: Ultrasound-guided Combined Pericapsular Nerve Group Block — With supine position, the probe will be put in a transverse plane along the anterior inferior iliac spine (AIIS) to identify the iliopsoas muscle, femoral nerve, and femoral artery (FA).
  Then the probe will be rotated counter clockwise to align with the pubic ramus to visualize the AIIS, iliopsoas prominence (IPE), FA, iliopsoas, and iliopsoas notch.
  Under direct vision, a 22-gauge, 50-mm echo needle will be advanced in the lateral-medial plane between the psoas tendon and the pubic ramus until the needle tip touches the IPE. The needle will be withdrawn, and after negative aspiration, 1 ml/kg (Bupivacaine 0.25%) is injected
  Arms: Group B
Procedure: Ultrasound-guided Lateral Femoral Cutaneous Nerve Block — patient remains supine, and the transducer is parallel to the inguinal ligament. With the femoral artery and vein as guidance, the lateral part of the sartorius muscle and fascia lata is visualized. Approximately 3 cm inferior from this point, the branches of the lateral femoral cutaneous nerve are visualized in the hypoechoic fat-filled subfascial space between the sartorius muscle medially and the tensor fascia lata muscle laterally. A 22-gauge, 50-mm needle is inserted with in plane approach at a shallow angle to reach the area of the nerve and after negative aspiration, 0.1 ml/kg (Bupivacaine 0.25%) is injected.
  Arms: Group B
Drug: Fentanyl — patients will receive an induction dose at 1 mcg/kg. If the analgesia was inadequate in the form of increase in heart rate and or arterial blood pressure by more than 20% of baseline values during surgery, this warrants the administration of intravenous fentanyl (0.5µg/kg).
Drug: Morphine — If a FLACC pain Score is ≥ 4/10, the patient in the PACU will receive morphine (intravenous, 0.03 mg/kg), and the maximum allowed dose is 0.1mg/kg every 4 hours.
  Other Names: rescue analgesia
Drug: Acetaminophen — P atients will receive postoperative IV acetaminophen IV 10 mg/ kg q 6 hours

SUMMARY:
combined pericapsular nerve group PENG block and lateral femoral cutaneous nerve block may be effective in reducing post-operative pain after open hip surgery in children.

DETAILED DESCRIPTION:
All children will be assessed clinically, and investigations will be done to exclude the exclusion criteria mentioned above. Laboratory works needed: complete blood count (CBC), prothrombin time, concentration, partial thromboplastin time. Midazolam (0.5mg/kg) will be given orally to each child in both groups as a premedication half an hour before the procedure.

General anesthesia will be induced in a supine position under standard basic monitoring of vital signs with inhalational anesthetic using (100%) O2 + Sevoflurane.

Group C will receive caudal analgesia Bupivacaine 0.25% at a dose of 1 ml/kg. Group B will receive PENG block Bupivacaine 0.25% at a dose of 1 ml/kg and lateral femoral cutaneous nerve block Bubivacaine 0.25% at 0.1 ml/kg.

After receiving the block, a surgical incision will be done after 15 minutes. Continuous recording of heart rate and blood pressure will be carried out from the moment of injection at timely intervals intra-operative. Intra-operatively, an increase in hemodynamics in response to the skin incision by more than 30% from baseline values 5 min after intubation or thereafter is managed by intravenous administration of fentanyl 1 µg/kg to a maximum dose of 2 µg/kg. Postoperative pain assessment using the FLACC score will then follow for 24 hours.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) physical status I, II.
* Unilateral hip surgery.

Exclusion Criteria:

* Parents' refusal to participate in the study.
* Coagulopathy (i.e. Platelets ≤ 50,000 and/or INR> 1.5).
* Localized infection at the site of needle insertion.
* Known hypersensitivity or allergies to any of the used drugs.
* Bilateral hip surgery in the same session.

Ages: 1 Year to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 68 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2024-07 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
Time to first rescue analgesia | First 24 hours postoperative
  Time (minutes) to first need of rescue analgesia postoperative.

SECONDARY OUTCOMES:
Intraoperative hemodynamic parameters | intraoperative period
  systolic, diastolic, mean blood pressure (mmHg)
Intraoperative hemodynamic parameters | intraoperative period
  heart rate (bpm)
Total fentanyl consumption | intraoperative period
  total intraoperative consumed fentanyl (mg/kg)
Total morphine consumption | First 24 hours postoperative
  total postoperative consumed morphine (mg/kg)
Postoperative pain assessment FLACC | First 24 hours postoperative
  In the PACU, quality of analgesia was assessed every 15 minutes for the first hour then after 2, 4 ,6 ,12,18 and 24 hours postoperative using (face, legs, activity, and cry consolability scale) (FLACC) pain score

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University Hospitals, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No